CLINICAL TRIAL: NCT00647179
Title: Substrate Metabolism and Insulin Sensitivity in Acromegalic Patients Before and After Treatment
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MM-ISA-20070130; M-20070130
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Acromegaly; Excessive Growth Hormone Secretion; Insulin Resistance
Keywords: Acromegaly; Growth Hormone; Insulin resistance; Glucose tolerance; Body Composition; Substrate metabolism
MeSH Terms: conditions — Acromegaly; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, muscle samples, fat samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients recently diagnosed with acromegaly
  Interventions: Procedure: Transsphenoidal adenomectomy

INTERVENTIONS:
Procedure: Transsphenoidal adenomectomy — Surgery

SUMMARY:
The purpose of this study is to investigate the effects of chronic elevated growth hormone on metabolism and insulin sensitivity by studying acromegalic patients before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written consent
* Age between 18 and 70
* Recently diagnosed with acromegaly

Exclusion Criteria:

* NYHA 3
* Uncontrolled hypertension
* Known cerebrovascular disease
* Proliferative retinopatia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patiens recently diagnoses with acromegaly, recruited from the clinic
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-02; Primary Completion 2016-12-07 (Actual); Study Completion 2016-12-07 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | Before and after treatment

SECONDARY OUTCOMES:
QoL, body composition, intrahepatic and intramyocellular fat, substrate metabolism, Glucose tolerance | Before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jørgensen, Professor MD, Principal Investigator — Aarhus University Hospital, Department of Endocrinology
Locations (1):
- Department of Endocrinology, Aarhus University Hospital, Aarhus C, Aarhus, Denmark

REFERENCES:
- [Derived] Arlien-Soborg MC, Grondahl C, Baek A, Dal J, Madsen M, Hogild ML, Pedersen SB, Bjerre M, Jorgensen JOL. Fibroblast Activation Protein is a GH Target: A Prospective Study of Patients with Acromegaly Before and After Treatment. J Clin Endocrinol Metab. 2020 Jan 1;105(1):dgz033. doi: 10.1210/clinem/dgz033. PMID 31544947